CLINICAL TRIAL: NCT07260305
Title: A Phase I , Open Label, Multi-center Study to Assess the Safety and Tolerability of KGX101 Mono and Combo Therapy With Envafolimab in Advanced or Metastatic Solid Tumor Patients
Brief Title: A Phase I Study to Investigate the Safety and Tolerability of KGX101 Monotherapy and Combination Therapy With Envafolimab in Advanced or Metastatic Solid Tumor Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kangabio AUSTRALIA LTD PTY (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGX101ST102
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — envafolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- KGX101 monotherapy-Dose level 1 (Experimental)
  Interventions: Drug: KGX101 injection
- KGX101 monotherapy-Dose level 2 (Experimental)
  Interventions: Drug: KGX101 injection
- KGX101 monotherapy-Dose level 3 (Experimental)
  Interventions: Drug: KGX101 injection
- KGX101 monotherapy-Dose level 4 (Experimental)
  Interventions: Drug: KGX101 injection
- KGX101 monotherapy dose expansion (Experimental)
  Interventions: Drug: KGX101 injection
- KGX101 combo with Envafolimab-Dose level 1 (Experimental)
  Interventions: Drug: KGX101 injection; Drug: Envafolimab
- KGX101 combo with Envafolimab-Dose level 2 (Experimental)
  Interventions: Drug: KGX101 injection; Drug: Envafolimab
- KGX101 combo with Envafolimab-Dose level 3 (Experimental)
  Interventions: Drug: KGX101 injection; Drug: Envafolimab
- KGX101 combo with Envafolimab dose expansion (Experimental)
  Interventions: Drug: KGX101 injection; Drug: Envafolimab

INTERVENTIONS:
Drug: KGX101 injection — KGX101 is a heterodimeric IL-12 prodrug with the C-terminus of IL-12 fused with ADCC-impaired IgG1 Fc and the N-terminus of IL-12 masked using the IL-12 binding domains of IL-12Rβ1 and IL-12Rβ2. KGX101 injection is a sterile, white or white-like lyophilized powder, supplied at 4.0 mg/vial for single use.
Drug: Envafolimab — Envafolimab is a novel fusion protein of humanized anti-PD-L1 single domain antibody and human IgG1 Fc fragment formulated for subcutaneous injection.
  Arms: KGX101 combo with Envafolimab dose expansion; KGX101 combo with Envafolimab-Dose level 1; KGX101 combo with Envafolimab-Dose level 2; KGX101 combo with Envafolimab-Dose level 3

SUMMARY:
This is a phase I, open-label, multi-center, dose escalation and expansion study in advanced or metastatic solid tumor patients. The're are two goals set in this study: one is to explore the safety and tolerability of KGX101 when mono and combo with envafolimab in Chinese patients, the other is to determine recommended phase 2 dose of KGX101 mono and combo with envafolimab. Participants will: 1. Take drug KGX101 mono or combo with envafolimab every 3 weeks; 2. Visit the clinic for checkups and tests. Schedule will be about 6-8 times in the first month and then about every 3 weeks afterwards.

ELIGIBILITY:
Inclusion Criteria:

1. Any histologically or cytologically confirmed solid tumor malignancy that is locally advanced or metastatic and has failed standard of care, no further standard can be used, or standard of care is not fit;
2. Eastern cooperative oncology grous performance status of 0-1;
3. Has at least 1 measurable lesion per RECIST 1.1;
4. Has adequate organ and bone marrow function as per study which including hemoglobin > 90 g/L, platelet count >=100*10e9/L, absolute meutrophil count >=1.5*10e9/L;
5. Life expectancy of at least 3 months;
6. Provision of signed and dated written inform consent prior to any study-related procedures, sampling and analyses.

Exclusion Criteria:

1. Active known second malignancy except adequately treated basal cell carcinoma, squamous cell skin cancer, in situ cervical cancer, breast cancer;
2. Patients with primary CNS malignancies;
3. Evidence of severe or uncontrolled systemic diseases, including: active infection, hypertension, chronically unhealed wound or ulcers;
4. Active autoimmnue disease requiring systemic treatment in the last 2 years, or immunodefiency which is on immunosuppressive therapy, chronic systemic or enteric steroid therapy;
5. History of pneumonitis, interstitial lung disease which require steroids or has current pneumonitis/ interstitial lung disease;
6. Any unresolved toxicities from prior therapy greater than CTCAE 5.0 grade 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with adverse events | From baseline to 30 days after the last dose administration.
  AE will be collected to assess participants' safety after KGX101 monotherapy or combo with Envafolimab
Number of participants with dose limiting toxicities/DLT within DLT observation period | From Day1 after the first priming dose of KGX101 until 21 days post the first target dose ofKGX101
  DLT will be observed from start of the first priming dose of KGX101 until 21 days post the first target dose of KGX101
Number of participants with changes of clinical lab abnormalities | From screening until 90 days post the last dose administration
  Any changes in values of the clinical chemistry, hematology, coagulation and urinalysis will be evaluated
The maximum tolerated dose of KGX101 monotherapy and combination therapy with Envafolimab | From Day 1 post the first dosing until 21 days post the the first target dosing

SECONDARY OUTCOMES:
PK parameters: Maximum Concentration (Cmax) of total IL-12 | Part A: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose. Part B: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose.
  Part A- The PK schedule after the first and third target dose injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Other sample collection timepoints include: pre-dose of each priming dose, pre-dose of other target dose; Part B- The PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters: Time of maximum observed concentration (Tmax)of total IL-12 | Part A: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose. Part B: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose.
  Part A- The PK schedule after the first and third target dose injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Other sample collection timepoints include: pre-dose of each priming dose, pre-dose of other target dose; Part B- The PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters: Area under the curve (AUC) | Part A: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose. Part B: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose.
  Part A- The PK schedule after the first and third target dose injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Other sample collection timepoints include: pre-dose of each priming dose, pre-dose of other target dose; Part B- The PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters: Half- life (T1 /2) | Part A: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose. Part B: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose.
  Part A- The PK schedule after the first and third target dose injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Other sample collection timepoints include: pre-dose of each priming dose, pre-dose of other target dose; Part B- The PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters- Trough concentration (Ctrough) | Part A: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose. Part B: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose.
  Part A- The PK schedule after the first and third target dose injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Other sample collection timepoints include: pre-dose of each priming dose, pre-dose of other target dose; Part B- The PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters- Systemic clearance (CL) | Part A: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose. Part B: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose.
  Part A- The PK schedule after the first and third target dose injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Other sample collection timepoints include: pre-dose of each priming dose, pre-dose of other target dose; Part B- The PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
PK Parameters- Volume of distribution (Vd) | Part A: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose. Part B: From pre-dose of the first dose of KGX101 treatment until Day 1 of the last dose.
  Part A- The PK schedule after the first and third target dose injection of KGX101 are as follows: pre-dose, 0 h, 2, 6, 24, 48, 72, 168 and 336hr post dose. Other sample collection timepoints include: pre-dose of each priming dose, pre-dose of other target dose; Part B- The PK schedule after Envafoliamb: pre-dose (1st, 2nd, 3rd and 4th treatment) and 72h ±1 h post the 1st Envafolimab treatment.
Immunogenicity- Anti-drug antibody (ADA) | Part A: From pre-dose of the first dose of KGX101 treatment until 90 days afrer the last dose. Part B: From pre-dose of the first dose of KGX101 treatment until 90 days after the last dose.
  Samples will be collected to assess the immunogeniccity after each KGX101 treatment.
Number of participants with changes in the Overall Response (ORR) | From Day 1 after the first dose of KGX101 till survival follow-up every 90 days post the last treatment.
Progression free survival (PFS) per RECIST 1.1 | From Day 1 after the first dose of KGX101 till survival follow-up every 90 days post last treatment.
Overall survival | From Day 1 after the first dose of KGX101 till survival follow-up every 90 days post last treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Principal Investigator — Beijing Cancer Hopspital
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fudan university Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided